CLINICAL TRIAL: NCT04572763
Title: A Phase I/II Study of Copanlisib Plus Venetoclax for the Treatment of Relapsed/Refractory Diffuse Large B-cell Lymphoma
Brief Title: Copanlisib Plus Venetoclax in R/R DLBCL
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: AbbVie (Industry); Bayer (Industry)
Responsible Party: Principal Investigator, Jennifer Crombie, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-069
Record Dates: First submitted 2020-09-22; First posted 2020-10-01 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Diffuse Large B Cell Lymphoma; Relapsed Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma
Keywords: Diffuse Large B Cell Lymphoma; Relapsed Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — copanlisib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Copanlisib + Venetoclax (Experimental): Phase 1
  * Dose escalation will occur using a 3+3 design
  * Copanlisib will be administered IV on days 1, 8 and 15 in 28 day cycle
  * Venetoclax will be administered orally daily for each 28-day cycle. During cycle 1, a venetoclax dose ramp-up is performed in the outpatient setting
  Interventions: Drug: Copanlisib; Drug: Venetoclax
- Recommended phase II dose (RP2D) Copanlisib + Venetoclax (Experimental): Patients will be treated with copanlisib in combination with venetoclax, administered at the Recommended phase II dose (RP2D).
  Interventions: Drug: Copanlisib; Drug: Venetoclax

INTERVENTIONS:
Drug: Copanlisib — Intravenous infusion
  Other Names: Aliqopa
Drug: Venetoclax — Tablet taken orally
  Other Names: Venclexta

SUMMARY:
This research study is evaluating the combination of two drugs, copanlisib and venetoclax, as a possible treatment for trelapsed/refractory diffuse large B-cell lymphoma (DLBCL)

The names of the study drugs involved in this study are:

* Copanlisib
* Venetoclax

DETAILED DESCRIPTION:
This study is an open-label, multi-center, non-randomized phase I/II study of the combination treatment copanlisib + venetoclax in patients with relapsed/refractory (R/R) diffuse large B-cell lymphoma (DLBCL).

Phase I clinical trials test the safety of investigational drugs, and also try to define the appropriate dose of the investigational drugs to use for further studies. Phase II clinical trials test the safety and effectiveness of investigational drugs to learn whether the drugs work in treating a specific disease."Investigational" means that the drugs are being studied.

Copanlisib is an IV medication that is approved by the U.S. Food and Drug Administration (FDA) for the treatment of adult patients with relapsed follicular lymphoma who have received at least two prior therapies. Venetoclax is an oral medication that is approved by the U.S. FDA for the treatment of adult patients with chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) and certain patients with acute myeloid leukemia (AML). The FDA has not approved copablisib or venetoclax for the treatment of DLBCL or the combination of copanlisib and venetoclax as a treatment for any disease.

In the phase I portion of this study, the investigators are looking to determine the dose of venetoclax that is safe to give with copanlisib and to see what the side effects are of this combination.

In the phase II trial, the investigators will be determining how effective venetoclax and copanlisib are for the treatment of R/R DLBCL. Data from laboratory suggest that some subsets of DLBCL are enriched for mutations that make them sensitive to the combination of copanlisib plus venetoclax. This study will look at genetic changes in your cancer and determine if abnormalities in specific genes make these drugs more or less effective.

It is expected that about 48 people will take part in this research study.

Bayer, a pharmaceutical company, is supporting this research study by providing the study drug copanlisib and funding for this study. Abbvie, a pharmaceutical company, is supporting this research study by providing the study drug venetoclax and funding for this study.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of DLBCL according to the 2016 WHO classification. Patients with high-grade B-cell lymphoma with translocations of MYC and BCL-2 and/or BCL-6 are eligible
* Relapsed after autologous stem cell transplantation or chimeric antigen receptor (CAR) T-cell therapy or not a candidate for these therapies
* Willingness to undergo a pre-treatment biopsy. If considered unsafe to proceed with biopsy, archival tissue samples may be utilized after discussion with the PI. Archival samples performed within 90 days and without intervening therapy are also acceptable if they meet the criteria as specified in the laboratory manual.
* ECOG performance status < 2
* Age ≥ 18 years
* Patients must meet the following hematologic criteria at screening:

  * Absolute neutrophil count ≥1000 cells/mm3 (0.5 x 109/L), with no white-blood cell growth factor use for at least 7 days prior to screening.
  * Platelet count ≥75,000 cells/mm3 (75 x 109/L) or ≥50,000 cells/mm3 (50 x 109/L if documented disease involvement of the bone marrow), without platelet transfusion within 7 days of screening
  * Hemoglobin (Hb) ≥ 8 g/dL, without blood transfusion within 7 days of screening
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN (≤ 5 x ULN for patients with liver involvement by lymphoma)
* Lipase ≤ 1.5 x ULN
* Total bilirubin ≤ 1.5 x ULN (< 3 x ULN for patients with Gilbert's syndrome, patients with cholestasis due to compressive adenopathies of the hepatic hilum or documented liver involvement or with biliary obstruction due to lymphoma)
* Adequate renal function defined by serum creatinine ≤1.5 x ULN or creatinine clearance (by Cockroft-Gault) ≥ 50 ml/min
* Women of childbearing potential (WOCBP) and men must agree to use effective contraception when sexually active. This applies for the time period between signing of the informed consent form and 6 months for WOCBP and for men after the last administration of study treatment. A woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include but are not limited to hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for continuous 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. The investigator or a designated associate is requested to advise the patient how to achieve highly effective birth control, e.g. intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner, use of two forms of birth control, and sexual abstinence. The use of condoms by male patients is required unless the female partner is permanently sterile.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients receiving cancer therapy (i.e., chemotherapy, radiation therapy, immunotherapy, biologic therapy, hormonal therapy, surgery and/or tumor embolization) within 2 weeks of Cycle 1/Day 1 with the following exceptions:

  * Limited palliative radiation is allowed if completed > 1 week of C1D1
  * Systemic corticosteroid therapy at a daily dose higher than 15 mg prednisone is allowed until C1D1.
* Chronic systemic corticosteroid therapy at a daily dose higher than 15 mg prednisone or equivalent.
* History of other malignancies, except:

  * Malignancy treated medically or surgically with curative intent and with no known active disease present for ≥2 years before the first dose of study drug
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease.
  * Localized prostate cancer and low-risk prostate cancer on active surveillance
* Within three months of autologous stem cell transplantation at time of starting study treatment
* Within six months of allogeneic stem cell transplantation at time of starting study treatment or active graft vs. host disease requiring systemic treatment or prophylaxis within 6 weeks of starting study treatment
* Vaccinated with live, attenuated vaccines of any kind <4 weeks before first dose of study drug
* History of or active autoimmune disease requiring systemic immunosuppression
* Recent infection requiring intravenous antibiotics that was completed ≤7 days before the first dose of study drug, or any uncontrolled active systemic infection
* Patients with ongoing use of prophylactic antibiotics are eligible as long as there is no evidence of active infection and the antibiotic is not included on the list of prohibited medications
* Known bleeding disorders (eg, von Willebrand's disease) or hemophilia
* History of stroke or intracranial hemorrhage within 3 months prior to enrollment
* Known history of Human Immunodeficiency Virus (HIV) infection. All patients must be screened for HIV up to 28 days prior to study drug start using a blood test for HIV according to local regulations.
* Hepatitis B (HBV) or hepatitis C (HCV). All patients must be screened for HBV and HCV up to 28 days prior to study drug start. Patients positive for HBsAg or HBcAb will be eligible if they are negative for HBV-DNA, these patients should receive prophylactic antiviral therapy. Patients positive for anti-HCV antibody will be eligible if they are negative for HCV-RNA.
* CMV PCR positive at baseline
* Major surgery within 4 weeks of first dose of study drug
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety at undue risk
* Uncontrolled arrhythmia or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization
* Unable to swallow capsules or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel currently affecting absorption, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction
* History of or concurrent condition of interstitial lung disease of any severity and/or severely impaired lung function (as judged by the investigator)
* Concurrent diagnosis of pheochromocytoma
* Lactating or pregnant. Women of child bearing potential must have a pregnancy test prior performed a maximum of 7 days before the start of treatment, and a negative result must be documented
* Patients receiving any other anti-cancer study agents
* Known lymphomatous involvement of the central nervous system
* Seizure disorder requiring medication
* Patients who require warfarin or other vitamin K antagonists for anticoagulation (other anticoagulants are allowed after consultation with the overall study chair).
* Concurrent administration of medications or foods that are strong inhibitors or inducers of CYP3A, CYP3A substrates with NTI, and P-gp inhibitors taken within 7 days of starting study treatment.
* Herbal medications excluded within 7 days of starting study treatment
* Uncontrolled arterial hypertension despite optimal medical management
* Type 1 or type 2 diabetes mellitus with a HbA1c > 8.5%
* Known hypersensitivity to any of the test drugs, test drug classes, or excipients in the formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-09-08 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2026-07-29 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of venetoclax in combination with copanlisib (recommended phase II dose (RP2D) - Phase 1 | 28 Days up to 1 year
  The highest dose of the drug combination that does not cause unacceptable side effects as assessed by protocol-specified DLT criteria.
Overall response rate (ORR) - Phase II | 28 Days
  Defined as the partial response (PR) and complete response (CR) rate, according to the Lugano criteria.

SECONDARY OUTCOMES:
Partial response Rate (PR) | 28 Days
  Per Lugano criteria
Complete response Rate (CR) | 28 Days
  Per Lugano criteria
Duration of response (DOR) | Every 3 months to 1 year
  Legnth of time the patients respond to therapy
Progression-free survival (PFS) | Time from randomization (or registration) to the date of first documented progression or date of death from any cause, whichever comes first, for up to 5 years.
  The time from randomization (or registration) to progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation.
Overall survival (OS) | Time from randomization (or registration) to the date of death from any cause, assessed for up to 5 years.
  The time from randomization (or registration) to death due to any cause or censored at date last known alive.
Exome sequencing | Up to 1 year
  A genomic classifier will be applied to whole exome sequencing (WES) of DLBCL biopsy samples to determine genomic cluster.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Crombie, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - City of Hope Cancer Center, Duarte, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Siteman Cancer Center at Washington University, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu